CLINICAL TRIAL: NCT05568940
Title: Evaluating Tibolone Add-back in Patients With Endometriosis and Fibroids
Acronym: eTAPE
Status: Withdrawn | Type: Observational
Why Stopped: More critical projects were prioritized.
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Andrew Zakhari, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2023-9075
Record Dates: First submitted 2022-09-25; First posted 2022-10-06 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Endometriosis; Fibroids
Keywords: Tibolone; Add-back hormone replacement therapy; GnRH-agonist injection; menopausal hormone therapy; chemically-induced menopause
MeSH Terms: conditions — Endometriosis; Leiomyoma | interventions — tibolone; Tablets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pre-menopausal women >18 years old with endometriosis and/or uterine fibroids: GnRH-a depot (11.25mg IM x 1) and daily Tibolone 2.5mg orally once a day for 2-3 months.
  Interventions: Drug: Tibolone 2.5 Mg Oral Tablet

INTERVENTIONS:
Drug: Tibolone 2.5 Mg Oral Tablet — Tibolone oral therapy for 2-3 months: All participants will take a Tibolone 2.5 mg tablet orally daily, at the same time each day, following a scheduled, luteal-phase injection of leuprolide acetate 11.25mg intramuscular (IM).
  Other Names: Livial

SUMMARY:
While there are many medical options for managing endometriosis and fibroids, GnRH-agonist (GnRH-a) therapy remains a very common method of treating these complex conditions. Although this therapy is effective, it does come with significant menopausal side effects, such as hot flashes, sweating, mood changes, sleep disturbance, altered sex drive, decreased bone density, and vaginal and urinary symptoms.

In short, chemically-induced menopause (menopause triggered by GnRH-a injection) causes the same symptoms of natural menopause, but with a sudden onset in a generally young and active population. Low dose hormone add-back therapy is commonly used to lessen these side effects of GnRH-a use.

There are many menopausal hormone therapies (MHTs) used in menopausal women that can help, but few studies have directly evaluated the different options of treatment for women undergoing chemically-induced menopause. Tibolone is a menopausal hormone therapy (MHT) that stands out as a good option in the management of medical menopause in endometriosis patients because it may give fewer side effects than other alternatives and have a positive effect on mood and libido.

This study aims to see how effective Tibolone is as an add-back therapy in women who are hormonally suppressed with a GnRH-a. For this study, we will recruit pre-menopausal women over the age of 18 years old undergoing therapy with the GnRH-a Lupron.

DETAILED DESCRIPTION:
Endometriosis is a common condition affecting approximately one in ten women, with significant adverse effects on women's quality of life and reproductive health. While there are numerous medical options for managing pain symptoms and reducing lesion size, GnRH-a therapy remains a mainstay of treating this complex condition. Similarly, uterine fibroids can cause heavy bleeding with associated anemia, and bulk symptoms, which may require surgical management. These hormone-sensitive fibroids regress and bleeding subsides when treatment with GnRH-a is used. This generally young and otherwise healthy population undergoes suppression of the hypothalamic-pituitary-ovarian axis in order to manage symptoms of either endometriosis or fibroids, or both if present concomitantly.

The efficacy of GnRH-a therapy has been extensively demonstrated in the literature albeit at the cost of significant menopausal side effects such as vasomotor symptoms, mood changes, sleep disturbance, altered libido, decreased bone mineral density, and genitourinary symptoms. In short, chemically-induced menopause confers the validated symptoms of natural menopause, but with an abrupt onset in a generally young and active population.

Add-back therapy with low-dose hormonal preparations is commonly used to mitigate the unwanted but largely inevitable adverse effects of GnRH-a use. Theoretically, any menopausal hormone therapy (MHT) used in menopausal women could serve the purpose, however few studies have evaluated directly the differing options in this unique population. One MHT preparation that stands out as a valuable option in the management of medical menopause in endometriosis patients is Tibolone. Tibolone is a synthetic steroid prodrug with active metabolites that exhibit estrogenic, progestogenic, and androgenic activity.

Prior studies have demonstrated that add-back treatment with Tibolone significantly reduces bone mineral density loss and vasomotor symptoms that normally occur with GnRH-a treatment. In addition, Tibolone has been shown to cause significantly fewer bleeding and spotting episodes and less breast tenderness than combined hormone replacement therapy (HRT) preparations, and has also been shown to improve mood and libido in menopausal women, making it a unique and attractive option in younger women undergoing temporary, chemical menopause.

This is a prospective open-label observational cohort study. Pre-menopausal women over 18 years of age with known or suspected endometriosis or uterine fibroids who will be undergoing treatment with an injectable GnRH-agonist (leuprolide acetate) at the Royal Victoria Hospital (Glen site) will be recruited and screened for exclusion criteria. Consenting participants of the study will receive a phone call before their GnRH-a treatment to report menopausal symptoms and endometriosis symptoms in a baseline evaluation. After their GnRH-a treatment, participants will be contacted, by phone call, one, two and three months post treatment to be asked a standardized set of questions to evaluate relief of menopausal symptoms, control of endometriosis symptoms, as well as adherence to treatment, and side-effects. Add-back will commence one month after the initial injection of GnRH-a, such that the incidence of vasomotor symptoms and other side-effects of GnRH-a may be observed. In this way, this is a crossover study by design in which patients will serve as their own controls, before and after initiating add-back therapy with Tibolone. Participants will always reserve the right to commence Tibolone sooner than 1 month if they experience bothersome side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal woman over 18 years of age with known or suspected endometriosis and/or uterine fibroids
* Undergoing medical management of endometriosis with a depot injection of GnRH-a for 3 months
* Off all other hormonal medications for the period of this treatment
* With or without history of recent hormonal treatment for endometriosis
* Able to provide informed consent

Exclusion Criteria:

* Allergy or contraindication to GnRH-a therapy, tibolone, or any contraindications to estrogen or progestin replacement
* Any uncontrolled endocrinopathy (ex: Pituitary gland disorder, uncontrolled hypothyroidism, etc)
* Prior hysterectomy
* Menopausal status
* Pregnant or seeking pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pre-menopausal women over 18 years of age with known or suspected endometriosis and/or uterine fibroids who will undergo medical management of endometriosis with a depot injection of GnRH-a for 3 months
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Patient reported relief of menopausal symptoms | Baseline
  Patient reported relief of menopausal symptoms will be evaluated using the Menopause rating scale (MRS).
  The MRS is a validated 11-item health-related quality of life scale (HRQoL), that measures the presence and severity of menopausal symptoms.
Patient reported relief of menopausal symptoms | 1 month following injection
  Patient reported relief of menopausal symptoms will be evaluated using the Menopause rating scale (MRS).
  The MRS is a validated 11-item health-related quality of life scale (HRQoL), that measures the presence and severity of menopausal symptoms.
Patient reported relief of menopausal symptoms | 2 months following injection
  Patient reported relief of menopausal symptoms will be evaluated using the Menopause rating scale (MRS).
  The MRS is a validated 11-item health-related quality of life scale (HRQoL), that measures the presence and severity of menopausal symptoms.
Patient reported relief of menopausal symptoms | 3 months following injection
  Patient reported relief of menopausal symptoms will be evaluated using the Menopause rating scale (MRS).
  The MRS is a validated 11-item health-related quality of life scale (HRQoL), that measures the presence and severity of menopausal symptoms.
Patient reported sexual function | Baseline
  Patient reported relief of sexual dysfunction (a menopausal symptom) will be evaluated using the Abbreviated female sexual function index (AFSFI).
  The abbreviated FSFI is a validated 6-item self-report questionnaire designed to assess female sexual function, comprised of six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain.
Patient reported sexual function | 1 month following injection
  Patient reported relief of sexual dysfunction (a menopausal symptom) will be evaluated using the Abbreviated female sexual function index (AFSFI).
  The abbreviated FSFI is a validated 6-item self-report questionnaire designed to assess female sexual function, comprised of six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain.
Patient reported sexual function | 2 months following injection
  Patient reported relief of sexual dysfunction (a menopausal symptom) will be evaluated using the Abbreviated female sexual function index (AFSFI).
  The abbreviated FSFI is a validated 6-item self-report questionnaire designed to assess female sexual function, comprised of six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain.
Patient reported sexual function | 3 months following injection
  Patient reported relief of sexual dysfunction (a menopausal symptom) will be evaluated using the Abbreviated female sexual function index (AFSFI).
  The abbreviated FSFI is a validated 6-item self-report questionnaire designed to assess female sexual function, comprised of six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain.

SECONDARY OUTCOMES:
Control of endometriosis symptoms | Baseline
  Control of endometriosis symptoms will be evaluated using a modified Biberoglu & Behrman (B&B) scale. This is a validated scale that evaluates endometriosis pain by patient's self-assessment of three pain symptoms (dysmenorrhea, dyspareunia, and chronic pelvic pain).
Control of endometriosis symptoms | 1 month following injection
  Control of endometriosis symptoms will be evaluated using a modified Biberoglu & Behrman (B&B) scale. This is a validated scale that evaluates endometriosis pain by patient's self-assessment of three pain symptoms (dysmenorrhea, dyspareunia, and chronic pelvic pain).
Control of endometriosis symptoms | 2 months following injection
  Control of endometriosis symptoms will be evaluated using a modified Biberoglu & Behrman (B&B) scale. This is a validated scale that evaluates endometriosis pain by patient's self-assessment of three pain symptoms (dysmenorrhea, dyspareunia, and chronic pelvic pain).
Control of endometriosis symptoms | 3 months following injection
  Control of endometriosis symptoms will be evaluated using a modified Biberoglu & Behrman (B&B) scale. This is a validated scale that evaluates endometriosis pain by patient's self-assessment of three pain symptoms (dysmenorrhea, dyspareunia, and chronic pelvic pain).
Tolerability of the regimen | 1 month following injection
  This will be discussed during the monthly phone call with the participant.
Tolerability of the regimen | 2 months following injection
  This will be discussed during the monthly phone call with the participant.
Tolerability of the regimen | 3 months following injection
  This will be discussed during the monthly phone call with the participant.
Incidence of major side effects | 1 month following injection
  This will be discussed during the monthly phone call with the participant.
Incidence of major side effects | 2 months following injection
  This will be discussed during the monthly phone call with the participant.
Incidence of major side effects | 3 months following injection
  This will be discussed during the monthly phone call with the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zakhari, M.D., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No